CLINICAL TRIAL: NCT05769712
Title: A Multicenter Cross-sectional Study of Shear Wave Ultrasound Imaging in Evaluating Supraspinatus Tendon Elasticity.
Acronym: SWE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Second Provincial General Hospital (Other)
Collaborators: The First Affiliated Hospital of Guangxi University of Chinese Medicine (Unknown); The People's Hospital of Chongzuo (Unknown); Dongguan People's Hospital (Other Government); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Dongguan Tungwah Hospital (Other); Yangjiang People's Hospital (Other); Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Tong Wang, physician, Guangdong Second Provincial General Hospital
Other Study IDs: Guangdong2ndcsk
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: supraspinatus tendon; Shear wave elastic imaging; ultrasound
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy people: Inclusion criteria：① Age range (above 18 years old); ② Non-professional athletes; ③ No medical history of shoulder and neck pain; ④ Ultrasound examination (-).
  Exclusion criteria: ① pregnant women or postpartum 1 year; ② Shoulder pain with active or passive cervical motion; ③ History of upper extremity trauma; (4) Shoulder surgery or treatment history, intra-articular injection history, use history of glucocorticoids, estrogens, quinolones and cholesterol drugs; (5) Shoulder joint fear test (shoulder joint abduction 90°, slowly increasing external rotation, the subject had a positive expression of fear); (6) Evidence of adhesive shoulder joint bursitis, such as the passive range of motion of the 2 motion planes of the shoulder joint is obviously limited; ⑦ Systemic autoimmune diseases, metabolic diseases, endocrine diseases, psoriasis; ⑧ unable to complete the relevant movements and positions; ⑨ Those who are reluctant to continue the experiment and ask to quit.
  Interventions: Diagnostic Test: Shear wave ultrasonic imaging
- diabetic: Inclusion criteria：① Age range (above 18 years old); ② Non-professional athletes; (3) Patients who meet the clinical guidelines for diabetes diagnosis and treatment and are diagnosed with diabetes (ADA guidelines 2020: patients with typical diabetes symptoms and random blood glucose ≥11.1 mmol/L or fasting blood glucose ≥7.0 mmol/L or 2h blood glucose ≥11.1 mmol/L after glucose loading without typical diabetes symptoms); ④ Medical history ≥2 years.
  Exclusion criteria: as above.
  Interventions: Diagnostic Test: Shear wave ultrasonic imaging

INTERVENTIONS:
Diagnostic Test: Shear wave ultrasonic imaging — Shear wave ultrasonic imaging technique was used to measure the superficial and deep shear wave velocity of supraspinatus tendon at 10mm (distal end) and 15mm (proximal end) from the attachment end of the greater tubercle of the humerus on the long axis section of supraspinatus tendon.

SUMMARY:
The goal of this multi-center, cross-sectional, observational study is to test and compare the difference of the supraspinatus tendon's elasticity between diabetics and healthy people. The main questions it aims to answer are:

* Ultrasonic characteristics of supraspinatus tendon in diabetic patients
* Influencing factors of elastic value and thickness of supraspinatus tendon

Participants will be asked to:

* Perform ultrasound examination of the shoulder join.
* Fill in a survey with certain questions on their basic information.

ELIGIBILITY:
Inclusion Criteria:

① Age range (above 18 years old); ② Non-professional athletes; ③ No medical history of shoulder and neck pain; ④ Ultrasound examination (-).

Exclusion criteria:

① pregnant women or postpartum 1 year; ② Shoulder pain with active or passive cervical motion; ③ History of upper extremity trauma; (4) Shoulder surgery or treatment history, intra-articular injection history, use history of glucocorticoids, estrogens, quinolones and cholesterol drugs; (5) Shoulder joint fear test (shoulder joint abduction 90°, slowly increasing external rotation, the subject had a positive expression of fear); (6) Evidence of adhesive shoulder joint bursitis, such as the passive range of motion of the 2 motion planes of the shoulder joint is obviously limited; ⑦ Systemic autoimmune diseases, metabolic diseases, endocrine diseases, psoriasis; ⑧ unable to complete the relevant movements and positions; ⑨ Those who are reluctant to continue the experiment and ask to quit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetic Inclusion criteria：① Age range (above 18 years old); ② Non-professional athletes; (3) Patients who meet the clinical guidelines for diabetes diagnosis and treatment and are diagnosed with diabetes (ADA guidelines 2020: patients with typical diabetes symptoms and random blood glucose ≥11.1 mmol/L or fasting blood glucose ≥7.0 mmol/L or 2h blood glucose ≥11.1 mmol/L after glucose loading without typical diabetes symptoms); ④ Medical history ≥2 years.
  Exclusion criteria: as above.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-11-05 (Estimated); Study Completion 2023-11-05 (Estimated)

PRIMARY OUTCOMES:
Elasticity of the supraspinatus tendon | 10 mins
  After activating the SWE mode, the elastic image was generated in the two-amplitude mode. After the image quality mode was qualified (the color curve in the figure was smooth), Shear wave velocity in the superficial and deep layers of the supraspinatus tendon were measured at the distal and proximal ends of the tendon perpendicular to the surface of the humerus, respectively.

SECONDARY OUTCOMES:
Thickness of the supraspinatus tendon | 2 mins
  The thickness of the supraspinatus tendon was measured at a tangent line perpendicular to the surface of the humerus 15mm from insertion.

OTHER OUTCOMES:
Blood flow within the supraspinatus tendon | 3 mins
  After activating the blood flow mode, the blood flow signal grading in the supraspinatus tendon was evaluated after the blood flow filled and stabilized.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong second provincial general hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breda SJ, van der Vlist A, de Vos RJ, Krestin GP, Oei EHG. The association between patellar tendon stiffness measured with shear-wave elastography and patellar tendinopathy-a case-control study. Eur Radiol. 2020 Nov;30(11):5942-5951. doi: 10.1007/s00330-020-06952-0. Epub 2020 Jun 4. PMID 32500197
- [Background] Abate M, Schiavone C, Salini V. Sonographic evaluation of the shoulder in asymptomatic elderly subjects with diabetes. BMC Musculoskelet Disord. 2010 Dec 7;11:278. doi: 10.1186/1471-2474-11-278. PMID 21138564
- [Background] Evranos B, Idilman I, Ipek A, Polat SB, Cakir B, Ersoy R. Real-time sonoelastography and ultrasound evaluation of the Achilles tendon in patients with diabetes with or without foot ulcers: a cross sectional study. J Diabetes Complications. 2015 Nov-Dec;29(8):1124-9. doi: 10.1016/j.jdiacomp.2015.08.012. Epub 2015 Aug 20. PMID 26382616
- [Background] Guney A, Vatansever F, Karaman I, Kafadar IH, Oner M, Turk CY. Biomechanical properties of Achilles tendon in diabetic vs. non-diabetic patients. Exp Clin Endocrinol Diabetes. 2015 Jul;123(7):428-32. doi: 10.1055/s-0035-1549889. Epub 2015 Apr 28. PMID 25918879
- [Background] Rosskopf AB, Ehrmann C, Buck FM, Gerber C, Fluck M, Pfirrmann CW. Quantitative Shear-Wave US Elastography of the Supraspinatus Muscle: Reliability of the Method and Relation to Tendon Integrity and Muscle Quality. Radiology. 2016 Feb;278(2):465-74. doi: 10.1148/radiol.2015150908. Epub 2015 Nov 5. PMID 26540450
- [Background] Lin DJ, Burke CJ, Abiri B, Babb JS, Adler RS. Supraspinatus muscle shear wave elastography (SWE): detection of biomechanical differences with varying tendon quality prior to gray-scale morphologic changes. Skeletal Radiol. 2020 May;49(5):731-738. doi: 10.1007/s00256-019-03334-6. Epub 2019 Dec 6. PMID 31811348